CLINICAL TRIAL: NCT07407894
Title: VITAL-Age Trial (iVS-1 Investigation for Targeting Aging and Longevity)
Brief Title: iVS-1 Probiotic Intervention Targeting Biological Aging in Midlife Adults
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synbiotic Health (Industry)
Collaborators: MusB Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MB-VITAL
Record Dates: First submitted 2026-01-28; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy Aging; Anti Aging
Keywords: Bifidobacterium adolescentis; iVS-1; Aging; Geroscience; Gut Microbiome; Probiotic; Healthspan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium adolescentis iVS-1 (Experimental): Probiotic Capsule
  Interventions: Dietary Supplement: Bifidobacterium adolescentis iVS-1
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium adolescentis iVS-1 — B. adolescentis iVS-1 (probiotic capsule) delivered orally once daily at a minimum of 8 billion CFU/day
  Arms: Bifidobacterium adolescentis iVS-1
Dietary Supplement: Placebo — Placebo capsule delivered orally once daily
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effects of Bifidobacterium adolescentis (iVS-1) supplementation on biological aging markers, metabolic health, and functional health outcomes in midlife adults. The study explores whether modulation of aging-related biological pathways through the gut microbiome may influence health-related outcomes.

DETAILED DESCRIPTION:
Aging is associated with progressive physiological changes involving inflammation, cellular senescence, mitochondrial function, and alterations in the gut microbiome. Interventions targeting these biological processes may influence age-related health outcomes. The gut microbiome plays a central and modifiable role, influencing metabolic health, inflammation, neurocognitive outcomes, and systemic aging processes.

Reductions in Bifidobacterium adolescentis have been observed with aging and have been associated with metabolic and inflammatory changes. Preliminary studies suggest that supplementation with this species may affect biological pathways relevant to aging.

This study is a randomized, double-blind, placebo-controlled trial designed to evaluate the effects of Bifidobacterium adolescentis (iVS-1) supplementation in adults aged 40-75 years. Participants will be randomized to receive iVS-1 (≥8 billion CFU per capsule) or placebo once daily for 150 days. Blood- and stool-based assessments and questionnaires about cognition, sleep quality, and quality of life will be collected at baseline, mid-intervention, and end of study.

Changes in these measures will be used to assess the relationship between Bifidobacterium adolescentis iVS-1 supplementation and biological aging markers, metabolic health, and functional health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-75 years.
* BMI: 20-34.9 kg/m².
* Able and willing to sign informed consent and participate for the study duration.

Exclusion Criteria:

* Chronic disease history (liver, kidney, heart).
* Current pregnancy and/or lactating.
* Colonoscopy and/or its preparation within 4 weeks of screening.
* Those who intend to have children during study period.
* Current probiotic, prebiotics and/or metabolic-altering supplement use.
* Those who are unable to cooperate with investigators and testing.
* Known history of cancer and/or ongoing cancer treatments.
* Abuse of drugs, alcohol, tobacco, nicotine and other substances.
* History of cardiac diseases: atherosclerosis, heart failure, unstable angina, stable angina, etc., and chronic hypoxic disease: emphysema, pulmonary heart disease and others related.
* History of chronic and major GI disease (pancreatitis, IBS, and IBD) and intestinal surgeries.
* Type 1 or 2 diabetes mellitus.
* Poorly controlled chronic diseases (hypertension, hyperlipidemia) that are clinically unstable.
* Vulnerable groups, including clinically ill, mentally ill, cognitively impaired, minors, and illiterate etc.
* Significant weight loss (>20%) in prior one month.
* Conditions affecting safety or outcome integrity.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Biological Aging Biomarkers | Baseline to Day 150
  Changes in gene expression of biomarkers associated with biological aging, assessed by quantitative polymerase chain reaction (qPCR), compared between placebo and study product groups over the study duration, including stratified analyses based on Bifidobacterium abundance.

SECONDARY OUTCOMES:
Change in Phenotypic Age | Baseline to Day 150
  Changes in Phenotypic Age calculated as a single value from blood-based biomarkers (albumin, creatinine, glucose, C-reactive protein, lymphocyte count, mean cell volume, red cell distribution width, alkaline phosphatase, and white blood cell count) and chronological age compared between placebo and study product groups over the study duration, including stratified analyses based on Bifidobacterium abundance.
Change in Bifidobacterium adolescentis iVS-1 Abundance | Baseline to Day 150
  Changes in fecal Bifidobacterium adolescentis iVS-1 abundance, assessed by quantitative polymerase chain reaction (qPCR), compared between placebo and study product groups over the study duration, including stratified analyses based on Bifidobacterium abundance.
Change in Metabolic Health Parameters | Baseline to Day 150
  Changes in metabolic and lipid biomarkers compared between placebo and study product groups over the study duration, including stratified analyses based on Bifidobacterium abundance.
Change in Cognitive Function | Baseline to Day 150
  Changes in global and executive cognitive function assessed using validated cognitive assessments compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Sleep Quality | Baseline to Day 150
  Changes in sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Quality of Life | Baseline to Day 150
  Changes in quality-of-life scores assessed using the Short Form-36 Health Survey (SF-36) compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.

OTHER OUTCOMES:
Change in Gut Microbiota Composition | Baseline to Day 150
  Changes in gut microbiome composition and diversity assessed using metagenomic sequencing of fecal samples compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Gut Microbiota Function | Baseline to Day 150
  Changes in gut microbiome function assessed using metagenomic sequencing of fecal samples compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Fecal Metabolites | Baseline to Day 150
  Changes in fecal and plasma metabolites, including short-chain fatty acids (SCFAs), bile acids, and trimethylamine N-oxide (TMAO) compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Gut Permeability Markers | Baseline to Day 150
  Changes in gut permeability markers assessed using validated enzyme-linked immunosorbent assay (ELISA) techniques compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.
Change in Inflammatory Markers | Baseline to Day 150
  Changes in inflammatory markers assessed using validated enzyme-linked immunosorbent assay (ELISA) techniques compared across timepoints and between placebo and study product groups, including stratified analyses based on Bifidobacterium abundance.

CONTACTS AND LOCATIONS:
Locations (1):
- MusB Research LLC, New Port Richey, Florida, United States

IPD SHARING:
Plan to Share IPD: No